CLINICAL TRIAL: NCT04514367
Title: A Phase 2a Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous ANX005 in Subjects With, or at Risk for, Manifest Huntington's Disease
Brief Title: An Open Label Study of ANX005 in Subjects With, or at Risk for, Manifest Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX005-HD-01
Record Dates: First submitted 2020-07-27; First posted 2020-08-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: ANX005 administered for up to 22 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ANX005 (Experimental): IV
  Interventions: Drug: ANX005

INTERVENTIONS:
Drug: ANX005 — Intravenous Infusion

SUMMARY:
This study is a multi-center, open-label study of intravenous (IV) ANX005 in subjects with, or at risk for, manifest Huntington's Disease (HD).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of intravenous ANX005 administered for up to 22 weeks in subjects with, or at risk for, manifest Huntington's Disease.

Subjects will receive induction dosing of ANX005 administered by IV infusion on Days 1 and 5 or 6, followed by maintenance dosing every 2 weeks through Week 22, with follow up visits on Weeks 24, 28, and 36.

All subjects will be contacted (in clinic visit or phone call) 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of or at risk for Huntington's disease: Genetically confirmed disease by direct DNA testing, total CAG-Age Product (CAP) score > 400 and UHDRS independence score ≥ 80.
2. Able to walk independently and self-sufficient in basic activities of daily living (e.g. eating, dressing, bathing).
3. All HD concomitant medications stable.
4. If female, must be postmenopausal (no menses for at least 2 years without an alternative medical cause), surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or agree to use highly effective methods of contraception.
5. Males with a woman of childbearing potential partner must agree to use highly effective methods of contraception.
6. Previously vaccinated against encapsulated bacterial pathogens (Neisseria meningitidis, Haemophilus influenzae, and Streptococcus pneumoniae) or willing to undergo vaccination.
7. Able to tolerate EEG and lumbar puncture (LP) procedures.

Exclusion Criteria:

1. Be at risk of suicide or self-harm within the preceding 12 months.
2. Chorea and/or cognitive deficits severe enough to interfere with study assessments.
3. Subjects with body weight > 150 kg.
4. Clinically significant findings on the screening laboratory testing or physical examination that are not specific to HD and may interfere with the conduct of the study or the interpretation of the data or increase subject risk.
5. Signs and symptoms of, or a diagnosis consistent with a chronic autoimmune disorder and/or an ANA titer ≥ 1:160.
6. History of previous infusion reactions, sensitivities, allergic, or anaphylactic reactions to previous medications, environmental stimuli or other substances.
7. Use of an experimental agent within 60 days or five half-lives prior to Screening or anytime over the duration of this study.
8. Prior treatment with any monoclonal antibody.
9. Presence of an implanted deep brain stimulation device.
10. Any history of gene therapy, RNA or DNA targeted HD specific investigational agents such as antisense oligonucleotides, cell transplantation or any experimental brain surgery.
11. Brain and spinal pathology that may interfere with cerebrospinal fluid homeostasis and circulation, increases intracranial pressure (implanted shunt or catheter), malformations or tumor.
12. Contraindication to undergoing an LP.
13. Hypersensitivity to any of the excipients in the ANX005 drug product.
14. Clinically significant intercurrent illness, medical condition, or medical history (including neurological or mental illness, HIV, any active infection, including Hepatitis B or C) that would jeopardize the safety of the subject, limit participation, or compromise the interpretation of the data derived from the subject.
15. Any known genetic deficiencies of the complement-cascade system.
16. History of chronic oral or intravenous steroid use or immunosuppressant medication use.
17. Hemoglobin, bilirubin, or lactate dehydrogenase (LDH) values that are outside normal limits and clinically significant or suggestive of hemolytic anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intravenous ANX005 administered for up to 22 weeks in subjects with, or at risk for, manifest Huntington's Disease | Up to Week 36
  As measured by incidence of TEAEs, SAEs, AEs related to ANX005, SAEs related to ANX005, Grade 3 or higher AEs, Grade 3 or higher AEs related to ANX005, AEs leading to study or treatment discontinuation.
Pharmacokinetics (PK) of ANX005 | Up to Week 36
  As measured by ANX005 serum and cerebrospinal fluid concentrations
Pharmacodynamics (PD) effects of ANX005 | Up to Week 36
  As measured by C1q, C4a, and NfL levels in blood and/or cerebrospinal fluid concentrations

OTHER OUTCOMES:
Exploratory effects of ANX005 on measures of efficacy | Up to Week 36
  As measured by Unified Huntington's Disease Rating Scale '99 (UHDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hoehn, MD, Study Director — Annexon, Inc.
Locations (6):
- United States (6):
  - Annexon Investigational Site 02, Birmingham, Alabama
  - Annexon Investigational Site 03, Englewood, Colorado
  - Annexon Investigational Site 04, Washington D.C., District of Columbia
  - Annexon Investigational Site 07, Durham, North Carolina
  - Annexon Investigational Site 06, Cincinnati, Ohio
  - Annexon Investigational Site 08, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No